CLINICAL TRIAL: NCT06176443
Title: Impact of an Increased Restrictive Factor of One Anastomosis Gastric Bypass Using a "FundoRing" Fundoplication on Metabolic Outcomes in Type 2 Diabetes Mellitus: a Randomized Controlled Trial
Brief Title: Impact of an Increased Restrictive Factor of One Anastomosis Gastric Bypass on Metabolic Outcomes Type 2 Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Society of Bariatric and Metabolic Surgeons of Kazakhstan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2_DM_F.R. 2020_2024
Record Dates: First submitted 2023-12-09; First posted 2023-12-19 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Obesity, Morbid; Diabetes Mellitus, Type 2
Keywords: Obesity; Metabolic Surgery; FundoRing; One anastomosis gastric bypass; Fundoplication; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- One anastomosis gastric bypass with combined fundoplication (Experimental): One anastomosis gastric bypass with combined fundoplication "FundoRing"
  Interventions: Procedure: One anastomosis gastric bypass with combined fundoplication
- One anastomosis gastric bypass without combined fundoplication (Active Comparator): One anastomosis gastric bypass without combined fundoplication
  Interventions: Procedure: One anastomosis gastric bypass without combined fundoplication

INTERVENTIONS:
Procedure: One anastomosis gastric bypass with combined fundoplication — FundoRingOAGB
  Arms: One anastomosis gastric bypass with combined fundoplication
Procedure: One anastomosis gastric bypass without combined fundoplication — OAGB
  Arms: One anastomosis gastric bypass without combined fundoplication

SUMMARY:
The purpose of the study is to evaluate the effect of an increased restrictive factor of one gastric anastomosis (OAGB) using a "FundoRing" fundoplication on metabolic outcomes in type 2 diabetes mellitus. The randomized controlled trial compared two interventional procedures: one group - using the original fundoplication procedure to enhance the restrictive effect and another group without fundoplication in the standard version of the OAGB.

DETAILED DESCRIPTION:
The randomized controlled trial compared two interventional procedures: one group - using the original fundoplication procedure to enhance the restrictive effect and another group without fundoplication in the standard version of the OAGB.

The purpose of the study is to evaluate the effect of an increased restrictive factor of one gastric anastomosis (OAGB) using a "FundoRing" fundoplication on metabolic outcomes in type 2 diabetes mellitus.

The main hypothesis is that an increase in the restrictive effect will lead to an increase in the metabolic effect and an increase in its persistence over time.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-55 kg/m2
* Patients with Diabetes Mellitus, Type 2

Exclusion Criteria:

* BMI <25 and >55 kg/m2
* Patients without Diabetes Mellitus, Type 2
* History of surgery on the stomach
* Less than 18 or more than 60 years of age
* Psychiatric illness
* Patients unwilling or unable to provide informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2024-01-13 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Metabolic improvements of type 2 diabetes | Baseline, at 12, 24, 36 months after surgery
  Change % of Glycosylated Hemoglobin. A1C level is below 5.7% - full remisson, a level of 5.7% to 6.4% indicates partial remission , and a level of 6.5% or more indicates diabetes

SECONDARY OUTCOMES:
Change of body mass index | Baseline, at 12, 24, 36 months after surgery
  The measure is assessing a change of body mass index. Weight (kg) and height (cm) will be combined with the report of measurement by body mass index (BMI) kg/m2

CONTACTS AND LOCATIONS:
Overall Officials: Oral Ospanov, Professor, Principal Investigator — Society of Bariatric and Metabolic Surgeons of Kazakhstan" (SBMSK)
Locations (1):
- Oral Ospanov, Astana, Aqmola, Kazakhstan